CLINICAL TRIAL: NCT02059057
Title: Crossover From IDE Trial CLN0009, Lung Volume Reduction Coil Treatment in Patients With Emphysema (RENEW) Study, IDE G110066
Brief Title: LVRC IDE Crossover Study (Crossover From IDE Trial CLN0009)
Acronym: CROSSOVER
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: FDA approval of supplementation to IDE/protocol amendment to terminate subject long term follow up
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: PneumRx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN0016
Record Dates: First submitted 2014-02-06; First posted 2014-02-11 (Estimated); Results first posted 2018-09-25 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Emphysema
MeSH Terms: conditions — Emphysema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LVRC System (Experimental)
  Interventions: Device: LVRC System

INTERVENTIONS:
Device: LVRC System

SUMMARY:
Crossover study for patients who were randomized to the Control Group in CLN0009 (NCT01608490).

DETAILED DESCRIPTION:
Provide LVRC procedure to qualifying subjects who were enrolled as Control Subjects in and completed the Lung Volume Reduction Coil Treatment in Patients with Emphysema (RENEW) Study, CLN0009, and obtain safety and effectiveness data on these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Subject was enrolled as a Control Subject in and completed all required study assessments through the 12 month visit for the Lung Volume Reduction Coil Treatment in Patients with Emphysema (RENEW) Study, CLN0009.
2. Subject has post-bronchodilator FEV1 ≤45% predicted.
3. Subject has residual volume (RV) ≥175% predicted.
4. Subject has stopped smoking for at least 8 weeks prior to entering the study, as confirmed by a Cotinine test or other appropriate diagnostic test.
5. Subject has read, understood and signed the Informed Consent form.
6. Subject has received Pneumococcal and Influenza vaccinations consistent with local recommendations and/or policy.

Exclusion Criteria:

1. Subject has severe homogeneous emphysema as determined by the Core Radiology Lab
2. Subject has co-morbidities that may significantly reduce subject's ability to improve exercise capacity (e.g. severe arthritis, planned knee surgery) or baseline limitation on 6MWT is not due to dyspnea.
3. Subject has a change in FEV1 >20% (or, for subjects with pre-bronchodilator FEV1 below 1 L, a change of > 200 mL) post-bronchodilator, unless investigator can confirm by other means that subject does not have asthma.
4. Subject has DLCO <20% of predicted.
5. Subject has severe gas exchange abnormalities as defined by:

   PaCO2 >55 mm Hg PaO2 <45 mm Hg on room air (High altitude criterion: PaO2 <30 mm Hg)
6. Subject has a history of recurrent clinically significant respiratory infections, defined as 3 hospitalizations for respiratory infection during the year prior to enrollment.
7. Subject has severe pulmonary hypertension. If pulmonary hypertension is present, "severe" is defined by right ventricular systolic pressure >50 mm Hg via right heart catheterization and/or echocardiogram.
8. Subject has an inability to walk >140 meters (150 yards) in 6 minutes.
9. Subject has evidence of other severe disease (such as, but not limited to, lung cancer or renal failure), which in the judgment of the investigator may compromise survival of the subject for the duration of the study.
10. Subject is pregnant or lactating, or plans to become pregnant within the study timeframe.
11. Subject has an inability to tolerate bronchoscopy under moderate sedation or general anesthesia.
12. Subject has clinically significant bronchiectasis.
13. Subject has giant bullae >1/3 lung volume.
14. Subject has had previous LVR surgery, lung transplantation, lobectomy, LVR devices or other devices to treat COPD in either lung.
15. Subject has been involved in pulmonary drug or device studies within 30 days prior to this study, with the exception of the RENEW Study.
16. Subject is taking >20 mg prednisone (or equivalent dose of a similar steroid) daily.
17. Subject requires high level chronic immunomodulatory therapy to treat a moderate to severe chronic inflammatory autoimmune disorder.
18. Subject is on an antiplatelet agent (such as Plavix) or anticoagulant therapy (such as heparin or Coumadin) which cannot be stopped for seven (7) days prior to procedure.
19. Subject has a sensitivity or allergy to nitinol (nickel-titanium) or its constituent metals.
20. Subject has a known sensitivity to drugs required to perform bronchoscopy.
21. Subject has been diagnosed with alpha-1 antitrypsin deficiency (AATD).
22. Subject has any other disease, condition(s) or habit(s) that would interfere with completion of study and follow up assessments, would increase risks of bronchoscopy or assessments, or in the judgment of the investigator would potentially interfere with compliance to this study or would adversely affect study outcomes.

    -

Min Age: 36 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2019-07-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (20):
  - University of Alabama Lung Health Center, Birmingham, Alabama
  - Cedars Sinai Medical Center, Los Angeles, California
  - El Camino Hospital/Palo Alto Medical Foundation, Mountain View, California
  - Yale University School of Medicine - Yale New Haven Hospital, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - Northwestern University, Chicago, Illinois
  - Illinois Lung and Critical Care Institute, Peoria, Illinois
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - New York Presbyterian Columbia University Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - The Cleveland Clinic, Cleveland, Ohio
  - Temple, Philadelphia, Pennsylvania
  - Emphysema COPD Research Center, University of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Pulmonary, Critical Care & Sleep Medicine Consultants,PCCS/St. Luke's Episcopal Hospital, Houston, Texas
  - University of Texas Health Sciences Center at San Antonio, San Antonio, Texas
  - Franciscan Research Center, Tacoma, Washington
  - University of Wisconsin School of Medicine & Public Health, Madison, Wisconsin
- Institut Universitaire de Cardiologie et de Pneumologie de Quebec (IUCPQ), Québec, Canada
- France (2):
  - Centre Hospitalier Universitaire de Nice, Nice
  - CHU de Reims - Hopital Maison Blanche, Reims
- University Medical Center Groningen, Groningen, Netherlands
- Royal Brompton Hospital & Chelsea Westminster, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- LVRC System: The Lung Volume Reduction Coil System is an implantable device, delivered through a fiber-optic bronchoscope. This is a two part system that consists of 1) sterile Nitinol Coils and 2) a sterile, disposable, single-use (single-patient) Delivery System consisting of a Guidewire, Catheter, Cartridge, and Forceps.
  RePneu Lung Volume Reduction Coil System: The LVRC group will undergo two bronchoscopic sessions under general or moderate sedation. During the procedure, subjects will be treated with Coils according to the Instructions for Use.
Period: Overall Study
Arm/Group | LVRC System
Started | 102
Completed | 87
Not Completed | 15

BASELINE CHARACTERISTICS:
Arm/Group | LVRC System
Number analyzed (Participants) | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58
  Male | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 101
  Unknown or Not Reported | 0
Six Minute Walk Test (6MWT) [Mean (Standard Deviation); unit: meters] — Mean absolute change from baseline to12 months. The six-minute walk test (6MWT) measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes. The individual is allowed to self-pace and rest as needed as they traverse back and forth along a marked walkway.
  meters | 313.6 (82.0)
Forced Expiratory Volume in one second (FEV1) [Mean (Standard Deviation); unit: Liters] — The forced expiratory volume in one second (FEV1) measurement shows the amount of air a person can forcefully exhale in one second. Typically, lower FEV1 scores show more severe stages of lung disease. A positive change in FEV1 indicates improvement in lung function.
  Liters | 0.7 (0.2)
Residual Volume (RV) [Mean (Standard Deviation); unit: Liters] — Residual volume is the amount of air that remains in a person's lungs after fully exhaling. A decrease in residual volume indicates improvement in patients with higher residual volume measures.
  Liters | 5.2 (1.3)
St. George's Respiratory Questionnaire (SGRQ) [Mean (Standard Deviation); unit: units of a scale] — The SGRQ is designed to measure health impairment in patients with asthma and COPD.
  It consists of 50 items and has two parts: Part I (Symptoms): several scales; Part II (Activity and Impacts): dichotomous (true/false) except last question (4-point Likert scale)
  Scores range from 0 to 100, with higher scores indicating more limitations.
  A negative change in score indicates improvement, with a mean change of 4 points being the minimal important difference.
  units of a scale | 57.9 (15.6)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Six Minute Walk Test (6MWT)
Description: Mean absolute change from baseline to12 months. The six-minute walk test (6MWT) measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes. The individual is allowed to self-pace and rest as needed as they traverse back and forth along a marked walkway.
Time Frame: Change in Baseline to 12 months
Population: Only patients who had both baseline and 12 month data were analyzed. Missing values were not imputed.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | LVRC System
Number analyzed (Participants) | 80
meters | -22.9 (72.6)

2. Secondary Outcome: Mean Percent Change in Forced Expiratory Volume in One Second (FEV1)
Description: The forced expiratory volume in one second (FEV1) measurement shows the amount of air a person can forcefully exhale in one second. Typically, lower FEV1 scores show more severe stages of lung disease. A positive change in FEV1 indicates improvement in lung function.
Time Frame: Change in Baseline to 12 months
Population: Only patients who had both baseline and 12 month data were analyzed. Missing values were not imputed.
Measure: Mean (Standard Deviation); unit: % change
Groups:
- LVRC System: LVRC System
Arm/Group | LVRC System
Number analyzed (Participants) | 83
% change | 2.2 (21.1)

3. Secondary Outcome: Mean Change in Residual Volume (RV)
Description: Residual volume is the amount of air that remains in a person's lungs after fully exhaling. A decrease in residual volume indicates improvement in patients with higher residual volume measures.
Time Frame: Change in Baseline to 12 months
Population: Only patients who had both baseline and 12 month data were analyzed. Missing values were not imputed.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | LVRC System
Number analyzed (Participants) | 81
Liters | -0.3 (0.7)

4. Secondary Outcome: Mean Change in St. Georges Respiratory Questionnaire (SGRQ)
Description: Measure Description: The SGRQ is designed to measure health impairment in patients with asthma and COPD.
  It consists of 50 items and has two parts: Part I (Symptoms): several scales; Part II (Activity and Impacts): dichotomous (true/false) except last question (4-point Likert scale)
  Scores range from 0 to 100, with higher scores indicating more limitations.
  A negative change in score indicates improvement, with a mean change of 4 points being the minimal important difference.
Time Frame: Change in Baseline to 12 months
Population: Only patients who had both baseline and 12 month data were analyzed. Missing values were not imputed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LVRC System
Number analyzed (Participants) | 83
units on a scale | -4.8 (14.8)

ADVERSE EVENTS:
Time Frame: 12 months
Description: Crossover subjects who had been treated with at least one procedure or entered the procedure room comprise the safety population (n=101) and are included in the safety analyses for this clinical study report.
Arm/Group | LVRC System
All-Cause Mortality (participants affected / at risk) | 9/101
Serious Adverse Events (participants affected / at risk) | 56/101
Other Adverse Events (participants affected / at risk) | 97/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LVRC System (N=101)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1)
Aortic Valve Stenosis (Cardiac disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1)
Cor Pulmonale (Cardiac disorders) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 1 (1)
Coronary Artery Occlusion (Cardiac disorders) | 1 (1)
Supraventricular Tachycardia (Cardiac disorders) | 1 (1)
Diabetic Gastroparesis (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Megacolon (Gastrointestinal disorders) | 1 (1)
Medical Device Complication (General disorders) | 3 (3)
Non-Cardiac Chest Pain (General disorders) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Aspergillosis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Infective Exacerbation of COPD (Infections and infestations) | 1 (2)
Lower Respiratory Tract Infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 17 (20)
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 1 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neuropathy Peripheral (Nervous system disorders) | 1 (1)
Renal Failure Acute (Renal and urinary disorders) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 23 (29)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LVRC System (N=101)
Chest Discomfort (General disorders) | 15 (21)
Chest Pain (General disorders) | 9 (9)
Medical Device Complication (General disorders) | 8 (8)
Non-Cardiac Chest Pain (General disorders) | 11 (14)
Pneumonia (Infections and infestations) | 20 (25)
Back Pain (Musculoskeletal and connective tissue disorders) | 6 (6)
Headache (Nervous system disorders) | 9 (11)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 62 (110)
Cough (Respiratory, thoracic and mediastinal disorders) | 16 (23)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17 (21)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 58 (96)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 18 (26)
Bronchitis (Infections and infestations) | 9 (11)
Nasopharyngitis (Infections and infestations) | 5 (5)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 7 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-08-24): https://cdn.clinicaltrials.gov/large-docs/57/NCT02059057/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-07): https://cdn.clinicaltrials.gov/large-docs/57/NCT02059057/SAP_001.pdf